CLINICAL TRIAL: NCT02089373
Title: A Pilot Study on Usefulness of Probe-based Confocal Laser Endomicroscopy Targeted Gastric Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2013-0392
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

ARMS (2):
- Probe-based confocal laser endomicroscopy (Experimental)
  Interventions: Procedure: Probe-based confocal laser endomicroscopy
- White light endoscopy (Active Comparator)
  Interventions: Procedure: White light endoscopy

INTERVENTIONS:
Procedure: Probe-based confocal laser endomicroscopy — In this arm1, an investigator observes a cancerous lesion using white light endoscopy. In addition, contrast dye for confocal laser endomicorscopy (fluorescein sodium 0.1mL/kg) is administered. Then, the cancerous lesion is observed using probe-based confocal laser endomicroscopy. The biopsy would be done 5 times at the most suspcious parts of the cancerous lesion.
  Arms: Probe-based confocal laser endomicroscopy
Procedure: White light endoscopy — In this arm2, an invesigator observes a cancerous lesion using white light endoscopy. The biopsy would be done 5 times at the most suspicious parts of the cancerous lesion.
  Arms: White light endoscopy

SUMMARY:
The purpose of this study is to conduct a study on genetic pathology, obtaining of pure cancer tissues is mandatory. Although the endoscopy with biopsy has been a gold standard for diagnosing gastric cancer, percentage of cancer cells in biopsy samples is usually 30% or less. Recently, confocal laser endomicroscopy has been introduced for real-time histopathologic diagnosis in various cancers. The investigators aim to evaluate that biopsy using probe-based confocal laser endomicroscopy will increase the percentage of cancer cells in biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

1. Age, between 20 and 80
2. Initial-onset gastric cancer which would be treated with surgery

Exclusion Criteria:

1. Previous subtotal gastrectomy
2. Pregnancy or breast milk feeding
3. Active infection
4. Significant cardiopulmonary disease
5. Active hepatitis or severe hepatic dysfunction
6. Severe renal dysfunction
7. Severe bone marrow dysfunction
8. Severe neurologic or psychotic disorder

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The percentage of cancer cells in biopsy samples | After 3 days from the end of the endoscopic submucosal dissection
  The percentages of cancer cells in biopsy samples according to the method of endoscopic method, probe-based confocal laser endomicroscopy versus white light endosocpy

CONTACTS AND LOCATIONS:
Locations (1):
- Institutional Review Board in Severance Hospital, Seodaemun-gu, Seoul, South Korea